CLINICAL TRIAL: NCT03538054
Title: Dextromethorphan in Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jarred Younger, Associate Professor; Director of the Neuroinflammation, Pain and Fatigue Laboratory, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: F161018005
Record Dates: First submitted 2018-01-19; First posted 2018-05-25 (Actual); Results first posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will not know when they are taking placebo or the study medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextromethorphan (Experimental): Participant will take one dextromethorphan 10mg capsule in the morning and at night.
  Interventions: Drug: Dextromethorphan
- Placebo (Placebo Comparator): Participants will take one placebo capsule in the morning and at night.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan — (1)10 mg, by mouth, twice daily every 12 hours.
  Arms: Dextromethorphan
Drug: Placebo — 1 capsule, by mouth, twice daily every 12 hours.
  Arms: Placebo

SUMMARY:
The objective of this protocol is to evaluate if Dextromethorphan (DXM) reduces Fibromyalgia (FM) pain. DXM is a drug found in several over-the-counter products, including cough suppressants. The drug may reduce FM pain by suppressing inflammation in the central nervous system. The investigators will be observing the effects of DXM on daily self-reported pain measures in people with FM. If DXM reduces FM pain, it will provide important information about the nature of FM pathophysiology.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic, widespread pain syndrome. Individuals with FM frequently report body pain, fatigue, sleep issues, cognitive impairment, headaches, and other symptoms. The disease affects approximately 5% of women in the United States. Many of those patients suffer with decreased quality of life and loss of employment.

The precise pathological mechanism of FM is not yet understood, and there is no targeted treatment for the condition. One hypothesis of FM with prior scientific support is that pain is caused by abnormal inflammation of the brain. When microglia cells in the brain adopt an inflammatory state, they release chemicals that can cause neurons to increase the transmission of pain signals.

DXM has been used in previous research and demonstrated to suppress pain symptoms. When given at higher dosages (above 200mg), the medication acts as a dissociative agent. This dosage can reduce pain, but produces side-effects that can limit daily functioning. At lower dosages, however, DXM may reduce inflammatory aspects of chronic pain while not causing dissociative side effects.

In animal models, central inflammation can be reduced with intraperitoneal dosages of DXM of 0.1mg/kg. In an average U.S. woman, this dosage would translate to approximately 8mg. Because an oral versus intraperitoneal dosing route will be used, the dose will be raised to 10mg, administered twice a day (once in the morning and once at night). The investigator will examine the impact of 20mg total daily DXM on self-reported FM pain.

ELIGIBILITY:
Inclusion Criteria:

1. Severe chronic fatigue ≥6 consecutive months not due to ongoing exertion or other medical condition associated with fatigue;
2. Daily self-reported pain of at least 4 out of 10;

3. Meets American College of Rheumatology 2016 case definition criteria for FM;

4. Able to attend UAB for all scheduled appointments;

5. Can complete daily self-reports of pain and other symptoms for duration of project.

Exclusion Criteria:

1. Blood draw contraindicated or otherwise not able to be performed;
2. High-sensitivity C-reactive protein (HS-CRP) ≥ 10 mg/L;
3. Erythrocyte sedimentation rate (ESR) >60 mm/hr;
4. Positive rheumatoid factor;
5. Positive anti-nuclear antibody (ANA);
6. Abnormal thyroid stimulating hormone or free thyroxine;
7. Diagnosed rheumatologic or auto-immune condition;
8. Blood or clotting disorder;
9. Use of blood thinning medication;
10. Current use of MAOI
11. Daily consumption of grapefruit juice
12. Oral temperature >100˚F at baseline;
13. Febrile illness or use of antibiotics in the 4 weeks before study commencement;
14. Planned surgery or procedures during the study period, or operated on in the 4 weeks before study commencement;
15. Pregnant or planning on becoming pregnant within 6 months, or currently breastfeeding
16. Regular use of any anti-inflammatory medication (such as aspirin, ibuprofen, naproxen);
17. Baseline HADS (Hospital Anxiety and Depression Scale) depression subscale score of ≥16;
18. Current litigation or worker's compensation claim;
19. Current participation in another treatment trial;
20. Planned vaccination during the study period, or vaccinated in the 4 weeks before study commencement.

Ages: 23 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jarred W Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama of Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants attended the in-person screening visit and were enrolled into the study. Of the 27 enrolled, 19 met inclusion criteria and began the study protocol.
Groups:
- Placebo First, Then Dextromethorphan: All participants first completed a 2 week baseline where they did not receive any medication. They then completed a 5 week placebo condition where they took one inert capsule in the morning and one at night. Following the placebo phase, participants completed 10 weeks of the dextromethorphan condition where they took one 10mg dextromethorphan in the morning, one 10mg dextromethorphan capsule at night.
Period: Baseline Phase (2 Weeks)
Arm/Group | Placebo First, Then Dextromethorphan
Started | 19
Completed | 18
Not Completed | 1
Not completed — Physician Decision | 1
Period: Placebo Phase (5 Weeks)
Arm/Group | Placebo First, Then Dextromethorphan
Started | 18
Completed | 16
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Dextromethorphan Phase (10 Weeks)
Arm/Group | Placebo First, Then Dextromethorphan
Started | 16
Completed | 14
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants first completed a 5-week placebo condition where they took one inert capsule in the morning, and one at night. They then completed a 10-week dextromethorphan condition where they took one 10 mg dextromethorphan capsule in the morning, and one at night.
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.07 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants] — Per the eligibility criteria, only female participants were recruited for this study.
  Participants
    Female | 14
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Duration of fibromyalgia illness [Mean (Standard Deviation); unit: years] | 10.19 (6.90)
Fibromyalgia severity [Mean (Standard Deviation); unit: units on a scale] — Fibromyalgia severity is based on a score of 0-31 utilizing the American College of Rheumatology's criteria, where 0 = no fibromyalgia symptoms and 31 = high severity of fibromyalgia symptoms.
  units on a scale | 22.14 (3.76)
Widespread Pain Index score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-19 with higher scores indicating higher levels of pain.
  units on a scale | 13.79 (2.91)
Symptom Severity Scale score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-12 with higher scores indicating more severe fibromyalgia symptoms.
  units on a scale | 8.36 (2.10)

OUTCOME MEASURES:

1. Primary Outcome: Daily Self-reported Pain Severity
Description: Daily self-reported widespread pain severity, rated on a 0 - 100 scale (0 = no pain and 100 = worst pain possible). Participants' daily scores from the last 4 weeks of each condition (placebo and dextromethorphan) were summed and then averaged across the 4-week time period.
Time Frame: Daily over 4 weeks
Population: All 14 participants underwent both the Dextromethorphan and Placebo conditions (within-subjects comparisons).
Measure: Mean (Standard Deviation); unit: score/day
Arm/Group | Dextromethorphan | Placebo
Number analyzed (Participants) | 14 | 14
score/day | 41.09 (24.32) | 45.55 (24.69)
Statistical Analysis 1: Comparison: Dextromethorphan vs Placebo; Test type: Superiority; p = 0.146, GEE — The clinical threshold was p < 0.05, with no corrections for multiple comparisons; Outcome scores were mean-centered by participant, allowing analyses to reflect within-person changes rather than between-person differences; Slope = -5.065

2. Secondary Outcome: Daily Self-reported Physical Activity
Description: Self-reported daily activity, rated from 0 - 100 where 0 is less daily activity and 100 is the most amount of daily activity. Participants' daily scores from the last 4 weeks of each condition (placebo and dextromethorphan) were summed and then averaged across the 4-week time period.
Time Frame: Daily over 4 weeks
Population: All 14 participants underwent both the Dextromethorphan and Placebo conditions (within-subjects comparisons).
Measure: Mean (Standard Deviation); unit: score/day
Arm/Group | Dextromethorphan | Placebo
Number analyzed (Participants) | 14 | 14
score/day | 46.92 (19.79) | 50.10 (19.70)
Statistical Analysis 1: Comparison: Dextromethorphan vs Placebo; Test type: Superiority; p = 0.052, GEE — The clinical threshold was p < 0.05, with no corrections for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Slope = 4.221

3. Secondary Outcome: Patient Global Impression of Change
Description: Patient global impression of change (PGIC) measured on a seven point likert scale (1 = "no change" to 7 = "a great deal better"). PGIC's were not administered to participants. The PGIC was inadvertently left out of the lab visit packet. Since the PGIC was not administered, data was not collected for both arms/groups.
Time Frame: 20 weeks
Population: Scores for the PGIC secondary outcome were not available for analyses due to administrator error. PGIC's were not administered to participants. The PGIC was inadvertently left out of the lab visit packet. Since the PGIC was not administered, data was not collected for both arms/groups.
Arm/Group | Dextromethorphan | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout participants' study completion, 19 weeks.
Groups:
- Placebo: Participants took one placebo capsule in the morning and one at night for 5 weeks.
- Dextromethorphan: Participant took one 10 mg dextromethorphan capsule in the morning and one at night for 10 weeks.
Arm/Group | Placebo | Dextromethorphan
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 7/14 | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Dextromethorphan (N=14)
Anxiety (Nervous system disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cold/respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Elevated alkaline phosphatase (Endocrine disorders) | 0 (0) | 2 (2)
Elevated alanine aminotransferase (Endocrine disorders) | 0 (0) | 3 (3)
Elevated chloride (Endocrine disorders) | 0 (0) | 1 (1)
Eye redness (Eye disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastrointestinal upset (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hot flashes (Endocrine disorders) | 0 (0) | 2 (2)
Low alkaline phosphatase (Endocrine disorders) | 1 (1) | 0 (0)
Low alanine aminotransferase (Endocrine disorders) | 0 (0) | 1 (1)
Low aspartate aminotransferase (Endocrine disorders) | 1 (1) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Medication was tested in a small number of fibromyalgia (FM) patients, limiting generalizability. Length of DXM treatment was only 10 weeks, so it is unclear if the results are durable. We used a single-blind design that could have led to experimenter bias. We relied only on self-reported pain rather than using objective pain assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT03538054/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03538054/SAP_002.pdf